CLINICAL TRIAL: NCT02081885
Title: Therapeutic Efficacy of Tricalcium Phosphate and Chitosan as Bone Regenerator Versus Autologous Graft in Surgery for Mandibular Fracture
Brief Title: Tricalcium Phosphate and Chitosan as Bone Regenerator Versus Autologous Graft in Surgery for Mandibular Fracture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, PhD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Chitosan-2014-1
Record Dates: First submitted 2014-01-31; First posted 2014-03-07 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Mandibular Fractures
Keywords: Tricalcium phosphate; Chitosan; Grafting, Bone; Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures | interventions — tricalcium phosphate; Chitosan; Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tricalcium Phosphate / Chitosan (Experimental)
  Interventions: Procedure: Tricalcium Phosphate / Chitosan
- Autologous Graft (Active Comparator)
  Interventions: Procedure: Autologous Graft

INTERVENTIONS:
Procedure: Tricalcium Phosphate / Chitosan
  Arms: Tricalcium Phosphate / Chitosan
Procedure: Autologous Graft
  Arms: Autologous Graft

SUMMARY:
Introduction After a mandibular fracture where bone has been lost, a number of complications and challenges are presented in trying to solve them. These defects are mainly classified into two groups: functional and cosmetic. The functional defects are incompetence of the lower lip, salivary incontinence, severe difficulty chewing and swallowing, temporomandibular joint disorders and difficulty in pronouncing words.

Esthetically facial asymmetry is produced with collapse of the affected side. Unreconstructed jaw retrusion and tends to offset the affected side, there is a change in mandibular movements, which, previous vertical movements are replaced by oblique or diagonal movements controlled by a single temporomandibular joint. It also presents a limitation in motility and lingual force, besides proprioception disorder left by the inferior alveolar nerve The loss of bone in mandibular fractures, is one of the great challenges facing maxillofacial surgery and unfortunately increasingly common. That's why they have done and are still doing research for the development of biomaterials, all with the purpose of trying to solve this problem by offering the patient better results than those obtained in the past, restoring both function and facial aesthetics according to each case

DETAILED DESCRIPTION:
Objective To evaluate the therapeutic efficacy of the combination of tricalcium phosphate and chitosan in comparison with autologous bone graft in bone regeneration applied to surgical mandibular fracture

Material and Methods Type of Study: Clinical Trial (Randomized) controlled This project will be performed in patients from the Service of Plastic and Reconstructive Surgery, Maxillofacial, Civil Hospital of Guadalajara Fray Antonio Alcalde diagnosed with facial fractures Computed tomography imaging study with axial and coronal skull, as well as three-dimensional reconstruction was performed, to obtain the size of the bone defect

Procedure A compound, with 5 grams of chitosan in an acidic solution, consisting of 2 ml acetic acid 99% water, is prepared. Leaving it under constant stirring for over 12 hours to obtain a chitosan acidic gel. The total volume of compound of chitosan will be doubly filtered to remove impurities and microorganisms that may contaminate the solution. The first filtration was carried out with Whatman paper No. 1 to remove residual impurities and the second whit nitrocellulose filter of 0.45 microns to ensure complete removal of bacteria and impurities. Once filtered, the chitosan compound be mixed with 0.2 g of tricalcium phosphate gauge and dispensed in 15-20ml in petri dishes and incubated at dry heat stove at 40 ° C for 16 hours or until completely evaporate the liquid phase, dehydration of the compound obtained in a thin film. The films of tricalcium phosphate and chitosan will be neutralized with 0.5% NaOH until evolution of the petri dish and then washed thoroughly with distilled water to remove traces of NaOH 0.5%. The film neutralized will be placed in a container for shape and incubated for 2 hours at 50 °C for drying. Subsequently, the films will be trimmed and sterilized in ultraviolet imager for 15 minutes and then sealed in packages of manufacturing list for your own use.

Description of the technical surgical To the patients selected for the protocol will be following the next described procedure; Under general inhaled anesthesia naso-tracheal via, we will proceed to clean with an adequate asepsis and antisepsis intraoral and face technique, sterile fields will be placed on a regular basis, and they will be infiltrate with lidocaine and epinephrine on the incision line depending on the type of approach. After this they will be incision in the skin and subcutaneous tissue, subsequently, with blunt dissection in deep planes, dissection of superficial cervical fascia and muscle platysma neck, until find the fracture traces in the jaw bone (depending on the classification on the anatomic localization). There will be a reduction of the fracture with manual traction, and placing a rigid bone fixation with plates and screws of titanium, and at the same time using cooling steril physiological solution to avoid overheating of the bone (at this moment the surgical process is identical in the two groups) after the end of this process and have a strong jaw, is then replaced the missing bone segment, the group with autologous graft from the iliac crest, where will be oblique incision with guidance bottom and back to the iliac crest, 1 cm from the back of the spine and approximate length of 5 cm, previous insertions of the abdominal muscles and external oblique Internal, until reach the periosteum.

The results package- lateral femoral cutaneous nerve and the lateral femoral cutaneous nerve are the only structures that must not be damaged during the dissection.

A court is performed with an osteotome behind, approximately 2 cm from the edge of the ridge, producing a fracture of the cortical leaving exposed the cancellous bone. The tables are transected bone, by means of an osteotome behind, in order to obtain a type of cortical graft-medullary, with a diameter no greater than 2.5 cm, the bleeding will be assessed and if necessary materials shall be used hemostatic, finally, it was sewn by planes with vicryl 000 and skin with nylon in 0000 to the end will be placed sterile dressing.

In the case of patients who are included in the group of the biomaterial composed of tricalcium phosphate and chitosan previously obtained in the laboratory and sterilized, will come in predetermined diameter of 2.5 x 2.5 cm. This will be clipped and adapted to the bone defect allowing intimate contact between the bone and the biomaterial.

When the intervention has been made (autologous graft or biomaterial), the incision will be approached by planes with vicryl 000 and at the skin with Nylon 000 sub dermal continued suture. At the end a sterile bandage is going to be placed and the surgery will be completed.

Statistical Analysis Nominal variables were analyzed using percentage frequencies, X2 test or Fisher exact test. Numeric variables using Student's t test for independent samples and ANOVA with post hoc Scheffe test. U Mann Whitney and Kruskal Wallis tests will be used as long as data do not conform to normal distribution. All values of p <0.05 was considered statistically significant. The analysis is going to do by using the SPSS v 17 for Windows program.

ELIGIBILITY:
Inclusion Criteria:

* Patients ot the service of reconstructive and plastic surgery of the Civil Hospital in Guadalajara Fray Antonio Mayor, with a diagnosis of traumatic mandibular fracture with bone defect < 2.5 cm.
* Wishing to participate in the study

Exclusion Criteria:

* Patients who have undergone radiation therapy.
* Psychiatric Patients.
* Patients who have not signed informed consent.
* Patients with Diabetes
* Patients with alterations in bone metabolism
* Patients with kidney diseases
* Patients who receipt corticosteroids
* Patients with heart disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Bone density determination in regenerated bone. | 30 days after the procedure.
  Determined with computed tomography measure by using Hounsfield Units.
Bone density determination in regenerated bone. | 6 months after the procedure.
  Determined with computed tomography measure by using Hounsfield Units.

SECONDARY OUTCOMES:
Classification of mandibular fracture | One day before surgery
  They will be classified as Nasal, Maxilla-malar, Dentoalveolar, Mandibular and Lefort fracture.
Edema | Patients will be followed daily from the immediate postoperative period until discharge, an expected average of 3 days.
  Identifying the presence or absence of edema.
Postoperative infection. | Patients will be followed daily from the immediate postoperative period until discharge, an expected average of 3 days.
  Identifying the different possible infectious postoperative complications.
Defect Size | 30 days after the procedure.
  According to the millimeters of bone structures missed.
Edema | 8 days after procedure.
  Identifying the presence or absence of edema.
Edema | 30 days after procedure.
  Identifying the presence or absence of edema.
Edema | 6 months after procedure.
  Identifying the presence or absence of edema.
Postoperative infection. | 8 days after procedure.
  Identifying the different possible infectious postoperative complications.
Postoperative infection. | 30 days after procedure.
  Identifying the different possible infectious postoperative complications.
Postoperative infection. | 6 months after procedure
  Identifying the different possible infectious postoperative complications.
Defect Size | 6 months after the procedure.
  According to the millimeters of bone structures missed.

OTHER OUTCOMES:
Age | One day before surgery
  Completed years
Gender | One day before surgery
  Male or Female

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez-Ojeda, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Civil Hospital of Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico